CLINICAL TRIAL: NCT04964089
Title: A Prospective, Randomized, Double-masked, Active Comparator-controlled, Multi-center, Two-arm, Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal KSI-301 Compared With Intravitreal Aflibercept in Participants With Neovascular (Wet) Age-related Macular Degeneration (wAMD)
Brief Title: A Study to Evaluate the Efficacy and Safety of Intravitreal KSI-301 Compared With Intravitreal Aflibercept in Participants With Neovascular (Wet) Age-related Macular Degeneration (wAMD)
Acronym: DAYLIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kodiak Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS301P107
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: AMD; Wet AMD; neovascularization secondary to age-related macular degeneration; KSI-301; Aflibercept; Vascular endothelial growth factor; VEGF; Anti-VEGF; Antibody biopolymer conjugate; Macular Degeneration; wAMD; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Vision, Low; Kodiak
MeSH Terms: conditions — Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders; Vision, Low | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into one of two treatment arms: KSI-301 or aflibercept.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: For masking purposes, sham injections will be administered at every monthly visit if an active treatment is not administered. To preserve masking, two investigators are required for this study. The masked Investigator will be responsible for the examinations and safety assessments. The unmasked Investigator will perform the injections and post-treatment assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KSI-301 (Treatment Group A) (Experimental): Intravitreal injection of KSI-301 (5 mg) at Day 1 once every 4 weeks via intravitreal injection through Week 44.
  Interventions: Drug: KSI-301
- Aflibercept (Treatment Group B) (Active Comparator): Intravitreal injection of aflibercept (2 mg) once every 4 weeks for 3 monthly doses followed by intravitreal injection of aflibercept (2 mg) once every 8 weeks from Week 16 to Week 44. Sham injections will be administered at each monthly visit where an active treatment is not administered.
  Interventions: Drug: Aflibercept; Other: Sham Procedure

INTERVENTIONS:
Drug: KSI-301 — Intravitreal Injection
  Arms: KSI-301 (Treatment Group A)
Drug: Aflibercept — Intravitreal Injection
  Other Names: Eylea
  Arms: Aflibercept (Treatment Group B)
Other: Sham Procedure — The sham is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.
  Arms: Aflibercept (Treatment Group B)

SUMMARY:
This Phase 3 study will evaluate the efficacy and safety of KSI-301 compared to aflibercept, in participants with neovascular (wet) age-related macular degeneration (wAMD)

DETAILED DESCRIPTION:
This is a Phase 3, prospective, randomized, double-masked, two-arm, multi-center non-inferiority study evaluating the efficacy and safety of repeated intravitreal dosing of KSI-301 5 mg in participants with visual impairment due to treatment-naïve neovascular (wet) age-related macular degeneration (wAMD)

The primary endpoint will be assessed as an average of Weeks 40, 44, and 48; additional secondary endpoints for efficacy will be assessed by visit over time

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to participation in the study.
* Treatment-naïve choroidal neovascularization (CNV) secondary to AMD.
* BCVA ETDRS score between 83 and 25 letters, inclusive, in the Study Eye.
* Decrease in vision in the Study Eye determined by the Investigator to be primarily the result of wAMD.
* Other protocol-specified inclusion criteria may apply

Exclusion Criteria:

* BCVA of hand motion or worse in the non-Study Eye or non-physical presence of a non-Study Eye (i.e., monocular).
* Active or suspected ocular or periocular infection or inflammation.
* CNV secondary to other causes in the Study Eye.
* Any history or evidence of a concurrent ocular condition present in the Study Eye, that in the opinion of the Investigator could require either medical or surgical intervention or affect macular edema or alter visual acuity during the study.
* Uncontrolled glaucoma in the Study Eye.
* Significant media opacities, including cataract, in the Study Eye that might interfere with visual acuity, assessment of safety, OCT or fundus photography.
* Cataract in the Study Eye that in the judgment of the Investigator is expected to require surgical extraction within 12 months of screening.
* Women who are pregnant or lactating or intending to become pregnant during the study.
* Recent history (within the 6 months prior to screening) of myocardial infarction, stroke, transient ischemic attack, acute congestive heart failure or any acute coronary event.
* History of a medical condition that, in the judgment of the Investigator, would preclude scheduled study visits, completion of the study, or a safe administration of investigational product.
* Uncontrolled blood pressure defined as a systolic value ≥180 mmHg or diastolic value ≥100 mmHg while at rest.
* Other protocol-specified exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Velazquez-Martin, MD, Study Director — Kodiak Sciences Inc
Locations (66):
- United States (65):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Northwest Arkansas Retina Associates, Springdale, Arkansas
  - California Retina Consultants, Bakersfield, California
  - Eye Medical Center of Fresno, Fresno, California
  - Retina Consultants of Orange County, Fullerton, California
  - UCSD Jacobs Retina Center, La Jolla, California
  - Retina Associates of Orange County, Laguna Hills, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Consultants of San Diego, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group Inc, Sacramento, California
  - Orange County Retina Medical Group, Santa Ana, California
  - Colorado Retina Associates PC, Lakewood, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Health Center, Fort Myers, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Retina Associates of Florida, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Springfield Clinic LLP, Springfield, Illinois
  - Talley Eye, Evansville, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates PA, Lenexa, Kansas
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants PC, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - New England Retina Consultants, Springfield, Massachusetts
  - Vitreo Retinal Associates PC, Worcester, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Associated Retinal Consultants PC, Royal Oak, Michigan
  - Vitreoretinal Surgery PA, Edina, Minnesota
  - Sierra Eye Associates, Reno, Nevada
  - The Retina Center of New Jersey, Bloomfield, New Jersey
  - NJ Retina, Teaneck, New Jersey
  - Retina-Vitreous Surgeons of Central NY, Liverpool, New York
  - Retina Associates of Western NY, Rochester, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cole Eye Institute, Cleveland, Ohio
  - Retina Northwest, Portland, Oregon
  - Retina Consultants, LLC, Salem, Oregon
  - Cascade Medical Research Institute, Springfield, Oregon
  - MidAtlantic Retina, Philadelphia, Pennsylvania
  - Retina Research of Beaufort, Beaufort, South Carolina
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates PC, Knoxville, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, Houston, Texas
  - Retina Consultants of Texas-(Katy), Katy, Texas
  - Texas Retina Associates, Plano, Texas
  - Austin Retina Associates (Round Rock), Round Rock, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Texas - (Woodlands), The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Spokane Eye, Spokane, Washington
- Emanuelli Research & Development Center LLC, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 94 medical centers between June 2021 and April 2022. The first participant was enrolled on 23 June 2021 and the last on 07 April 2022.
Pre-assignment Details: Of 815 participants screened, 557 were randomized to treatment.
Period: Overall Study
Arm/Group | KSI-301 (Treatment Group A) | Aflibercept (Treatment Group B)
Started | 276 | 281
Completed | 253 | 268
Not Completed | 23 | 13
Not completed — Adverse Event | 8 | 6
Not completed — Non-compliance with study schedule | 1 | 0
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Progressive disease | 4 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Participant did not want to continue study treatment | 1 | 0
Not completed — Participant moved to different state | 1 | 0
Not completed — Participant decided to discontinue | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects who received at least one active study treatment (KSI-301 or aflibercept)
Groups:
- Total: Total of all reporting groups
Arm/Group | KSI-301 (Treatment Group A) | Aflibercept (Treatment Group B) | Total
Number analyzed (Participants) | 276 | 281 | 557
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 257 | 263 | 520
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.9 (8.21) | 77.2 (7.84) | 77.0 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 180 | 339
  Male | 117 | 101 | 218
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 14 | 30
  Not Hispanic or Latino | 260 | 267 | 527
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 2 | 0 | 2
  White | 269 | 276 | 545
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 1 | 1
Geographic Region [Count of Participants; unit: Participants]
  North America | 225 | 228 | 453
  Rest of World | 51 | 53 | 104
BCVA in the Study Eye [Mean (Standard Deviation); unit: Letters] | 63.7 (13.06) | 64.0 (13.09) | 63.8 (13.07)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) From Day 1 to the Average of Non-missing BCVA Values of Weeks 40, 44 and 48.
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity.
Time Frame: Day 1 to Week 48
Population: Full analysis set defined as all randomized subjects who received at least one treatment injection. Subjects will be analyzed according to their randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: ETDRS Letters
Arm/Group | KSI-301 (Treatment Group A) | Aflibercept (Treatment Group B)
Number analyzed (Participants) | 276 | 281
ETDRS Letters | 2.5 (0.78) | 4.6 (0.76)
Statistical Analysis 1: Comparison: KSI-301 (Treatment Group A) vs Aflibercept (Treatment Group B); Test type: Non-Inferiority — The maximum clinically acceptable true difference between KSI-301 and aflibercept participants to be considered non-inferior is 4.5 ETDRS letters, i.e. the non-inferiority margin (NI) is 4.5 letters; p = 0.0083, Mixed Models Analysis; MMRM model with treatment, visit, treatment by visit interaction, randomization stratification factors, and continuous baseline BCVA as covariates; Adjusted mean difference = -2.1, 95.03% CI 2-sided [-3.88 to -0.29], Standard Error of Mean 0.91

2. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) by Visit Over Time
Description: as for outcome 1
Time Frame: Day 1 to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | KSI-301 (Treatment Group A) | Aflibercept (Treatment Group B)
Number analyzed (Participants) | 276 | 281
ETDRS Letters
  Week 2: number analyzed (Participants) | 270 | 275
  Week 2 | 2.8 (6.48) | 2.9 (7.12)
  Week 4: number analyzed (Participants) | 273 | 278
  Week 4 | 3.4 (7.05) | 4.2 (7.29)
  Week 8: number analyzed (Participants) | 274 | 274
  Week 8 | 3.7 (8.52) | 5.1 (7.86)
  Week 12: number analyzed (Participants) | 267 | 274
  Week 12 | 3.8 (8.83) | 5.4 (7.90)
  Week 16: number analyzed (Participants) | 264 | 274
  Week 16 | 3.6 (9.09) | 4.9 (8.54)
  Week 20: number analyzed (Participants) | 262 | 275
  Week 20 | 3.9 (9.60) | 5.7 (8.97)
  Week 24: number analyzed (Participants) | 261 | 270
  Week 24 | 4.5 (9.29) | 6.0 (9.45)
  Week 28: number analyzed (Participants) | 257 | 263
  Week 28 | 4.5 (9.75) | 6.1 (9.49)
  Week 32: number analyzed (Participants) | 252 | 268
  Week 32 | 3.9 (10.32) | 6.1 (9.86)
  Week 36: number analyzed (Participants) | 250 | 266
  Week 36 | 3.7 (10.58) | 6.1 (9.77)
  Week 40: number analyzed (Participants) | 246 | 265
  Week 40 | 4.0 (11.05) | 5.6 (10.75)
  Week 44: number analyzed (Participants) | 240 | 260
  Week 44 | 4.7 (9.99) | 5.9 (10.71)
  Week 48: number analyzed (Participants) | 245 | 262
  Week 48 | 3.7 (11.12) | 5.4 (11.36)

3. Secondary Outcome: Proportion of Patients Who Gain ≥ 5, ≥10 and ≥15 Letters From Baseline Over Time
Description: Categorical improvements in Best Corrected Visual Acuity (BCVA) of clinically relevant BCVA measurements corresponding to 1, 2 and 3 lines of the ETDRS vision testing chart
Time Frame: Day 1 to Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Treatment Group A) | Aflibercept (Treatment Group B)
Number analyzed (Participants) | 276 | 281
Participants
  Gain ≥5 ETDRS Letters at Week 2: number analyzed (Participants) | 270 | 275
  Gain ≥5 ETDRS Letters at Week 2 | 100 | 96
  Gain ≥5 ETDRS Letters at Week 4: number analyzed (Participants) | 273 | 278
  Gain ≥5 ETDRS Letters at Week 4 | 110 | 129
  Gain ≥5 ETDRS Letters at Week 8: number analyzed (Participants) | 274 | 274
  Gain ≥5 ETDRS Letters at Week 8 | 119 | 151
  Gain ≥5 ETDRS Letters at Week 12: number analyzed (Participants) | 267 | 274
  Gain ≥5 ETDRS Letters at Week 12 | 124 | 148
  Gain ≥5 ETDRS Letters at Week 16: number analyzed (Participants) | 264 | 274
  Gain ≥5 ETDRS Letters at Week 16 | 119 | 143
  Gain ≥5 ETDRS Letters at Week 20: number analyzed (Participants) | 262 | 275
  Gain ≥5 ETDRS Letters at Week 20 | 121 | 161
  Gain ≥5 ETDRS Letters at Week 24: number analyzed (Participants) | 261 | 270
  Gain ≥5 ETDRS Letters at Week 24 | 130 | 156
  Gain ≥5 ETDRS Letters at Week 28: number analyzed (Participants) | 257 | 263
  Gain ≥5 ETDRS Letters at Week 28 | 122 | 154
  Gain ≥5 ETDRS Letters at Week 32: number analyzed (Participants) | 252 | 268
  Gain ≥5 ETDRS Letters at Week 32 | 132 | 168
  Gain ≥5 ETDRS Letters at Week 36: number analyzed (Participants) | 250 | 266
  Gain ≥5 ETDRS Letters at Week 36 | 120 | 158
  Gain ≥5 ETDRS Letters at Week 40: number analyzed (Participants) | 246 | 265
  Gain ≥5 ETDRS Letters at Week 40 | 116 | 156
  Gain ≥5 ETDRS Letters at Week 44: number analyzed (Participants) | 240 | 260
  Gain ≥5 ETDRS Letters at Week 44 | 126 | 151
  Gain ≥5 ETDRS Letters at Week 48: number analyzed (Participants) | 245 | 262
  Gain ≥5 ETDRS Letters at Week 48 | 111 | 150
  Gain ≥10 ETDRS Letters at Week 2: number analyzed (Participants) | 270 | 275
  Gain ≥10 ETDRS Letters at Week 2 | 31 | 37
  Gain ≥10 ETDRS Letters at Week 4: number analyzed (Participants) | 273 | 278
  Gain ≥10 ETDRS Letters at Week 4 | 44 | 54
  Gain ≥10 ETDRS Letters at Week 8: number analyzed (Participants) | 274 | 274
  Gain ≥10 ETDRS Letters at Week 8 | 52 | 72
  Gain ≥10 ETDRS Letters at Week 12: number analyzed (Participants) | 267 | 274
  Gain ≥10 ETDRS Letters at Week 12 | 55 | 72
  Gain ≥10 ETDRS Letters at Week 16: number analyzed (Participants) | 264 | 274
  Gain ≥10 ETDRS Letters at Week 16 | 62 | 68
  Gain ≥10 ETDRS Letters at Week 20: number analyzed (Participants) | 262 | 275
  Gain ≥10 ETDRS Letters at Week 20 | 66 | 86
  Gain ≥10 ETDRS Letters at Week 24: number analyzed (Participants) | 261 | 270
  Gain ≥10 ETDRS Letters at Week 24 | 70 | 90
  Gain ≥10 ETDRS Letters at Week 28: number analyzed (Participants) | 257 | 263
  Gain ≥10 ETDRS Letters at Week 28 | 66 | 87
  Gain ≥10 ETDRS Letters at Week 32: number analyzed (Participants) | 252 | 268
  Gain ≥10 ETDRS Letters at Week 32 | 57 | 95
  Gain ≥10 ETDRS Letters at Week 36: number analyzed (Participants) | 250 | 266
  Gain ≥10 ETDRS Letters at Week 36 | 66 | 81
  Gain ≥10 ETDRS Letters at Week 40: number analyzed (Participants) | 246 | 265
  Gain ≥10 ETDRS Letters at Week 40 | 67 | 80
  Gain ≥10 ETDRS Letters at Week 44: number analyzed (Participants) | 240 | 260
  Gain ≥10 ETDRS Letters at Week 44 | 67 | 86
  Gain ≥10 ETDRS Letters at Week 48: number analyzed (Participants) | 245 | 262
  Gain ≥10 ETDRS Letters at Week 48 | 65 | 85
  Gain ≥15 ETDRS Letters at Week 2: number analyzed (Participants) | 270 | 275
  Gain ≥15 ETDRS Letters at Week 2 | 12 | 11
  Gain ≥15 ETDRS Letters at Week 4: number analyzed (Participants) | 273 | 278
  Gain ≥15 ETDRS Letters at Week 4 | 18 | 21
  Gain ≥15 ETDRS Letters at Week 8: number analyzed (Participants) | 274 | 274
  Gain ≥15 ETDRS Letters at Week 8 | 24 | 28
  Gain ≥15 ETDRS Letters at Week 12: number analyzed (Participants) | 267 | 274
  Gain ≥15 ETDRS Letters at Week 12 | 20 | 29
  Gain ≥15 ETDRS Letters at Week 16: number analyzed (Participants) | 264 | 274
  Gain ≥15 ETDRS Letters at Week 16 | 24 | 33
  Gain ≥15 ETDRS Letters at Week 20: number analyzed (Participants) | 262 | 275
  Gain ≥15 ETDRS Letters at Week 20 | 28 | 33
  Gain ≥15 ETDRS Letters at Week 24: number analyzed (Participants) | 261 | 270
  Gain ≥15 ETDRS Letters at Week 24 | 33 | 42
  Gain ≥15 ETDRS Letters at Week 28: number analyzed (Participants) | 257 | 263
  Gain ≥15 ETDRS Letters at Week 28 | 36 | 46
  Gain ≥15 ETDRS Letters at Week 32: number analyzed (Participants) | 252 | 268
  Gain ≥15 ETDRS Letters at Week 32 | 32 | 37
  Gain ≥15 ETDRS Letters at Week 36: number analyzed (Participants) | 250 | 266
  Gain ≥15 ETDRS Letters at Week 36 | 32 | 44
  Gain ≥15 ETDRS Letters at Week 40: number analyzed (Participants) | 246 | 265
  Gain ≥15 ETDRS Letters at Week 40 | 33 | 45
  Gain ≥15 ETDRS Letters at Week 44: number analyzed (Participants) | 240 | 260
  Gain ≥15 ETDRS Letters at Week 44 | 34 | 48
  Gain ≥15 ETDRS Letters at Week 48: number analyzed (Participants) | 245 | 262
  Gain ≥15 ETDRS Letters at Week 48 | 35 | 49

4. Secondary Outcome: Proportion of Patients Who Lost ≥ 5, ≥10 and ≥15 Letters From Baseline Over Time
Description: Categorical worsening in Best Corrected Visual Acuity (BCVA) of clinically relevant BCVA measurements corresponding to 1, 2 and 3 lines of the ETDRS vision testing chart
Time Frame: Day 1 to Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Treatment Group A) | Aflibercept (Treatment Group B)
Number analyzed (Participants) | 276 | 281
Participants
  Loss ≥ 5 ETDRS Letters at Week 2: number analyzed (Participants) | 270 | 275
  Loss ≥ 5 ETDRS Letters at Week 2 | 20 | 28
  Loss ≥ 5 ETDRS Letters at Week 4: number analyzed (Participants) | 273 | 278
  Loss ≥ 5 ETDRS Letters at Week 4 | 27 | 19
  Loss ≥ 5 ETDRS Letters at Week 8: number analyzed (Participants) | 274 | 274
  Loss ≥ 5 ETDRS Letters at Week 8 | 41 | 22
  Loss ≥ 5 ETDRS Letters at Week 12: number analyzed (Participants) | 267 | 274
  Loss ≥ 5 ETDRS Letters at Week 12 | 35 | 24
  Loss ≥ 5 ETDRS Letters at Week 16: number analyzed (Participants) | 264 | 274
  Loss ≥ 5 ETDRS Letters at Week 16 | 35 | 31
  Loss ≥ 5 ETDRS Letters at Week 20: number analyzed (Participants) | 262 | 275
  Loss ≥ 5 ETDRS Letters at Week 20 | 35 | 27
  Loss ≥ 5 ETDRS Letters at Week 24: number analyzed (Participants) | 261 | 270
  Loss ≥ 5 ETDRS Letters at Week 24 | 34 | 31
  Loss ≥ 5 ETDRS Letters at Week 28: number analyzed (Participants) | 257 | 263
  Loss ≥ 5 ETDRS Letters at Week 28 | 38 | 31
  Loss ≥ 5 ETDRS Letters at Week 32: number analyzed (Participants) | 252 | 268
  Loss ≥ 5 ETDRS Letters at Week 32 | 41 | 35
  Loss ≥ 5 ETDRS Letters at Week 36: number analyzed (Participants) | 250 | 266
  Loss ≥ 5 ETDRS Letters at Week 36 | 47 | 32
  Loss ≥ 5 ETDRS Letters at Week 40: number analyzed (Participants) | 246 | 265
  Loss ≥ 5 ETDRS Letters at Week 40 | 33 | 41
  Loss ≥ 5 ETDRS Letters at Week 44: number analyzed (Participants) | 240 | 260
  Loss ≥ 5 ETDRS Letters at Week 44 | 33 | 33
  Loss ≥ 5 ETDRS Letters at Week 48: number analyzed (Participants) | 245 | 262
  Loss ≥ 5 ETDRS Letters at Week 48 | 39 | 38
  Loss ≥ 10 ETDRS Letters at Week 2: number analyzed (Participants) | 270 | 275
  Loss ≥ 10 ETDRS Letters at Week 2 | 6 | 10
  Loss ≥ 10 ETDRS Letters at Week 4: number analyzed (Participants) | 273 | 278
  Loss ≥ 10 ETDRS Letters at Week 4 | 6 | 4
  Loss ≥ 10 ETDRS Letters at Week 8: number analyzed (Participants) | 274 | 274
  Loss ≥ 10 ETDRS Letters at Week 8 | 10 | 8
  Loss ≥ 10 ETDRS Letters at Week 12: number analyzed (Participants) | 267 | 274
  Loss ≥ 10 ETDRS Letters at Week 12 | 15 | 9
  Loss ≥ 10 ETDRS Letters at Week 16: number analyzed (Participants) | 264 | 274
  Loss ≥ 10 ETDRS Letters at Week 16 | 15 | 15
  Loss ≥ 10 ETDRS Letters at Week 20: number analyzed (Participants) | 262 | 275
  Loss ≥ 10 ETDRS Letters at Week 20 | 16 | 14
  Loss ≥ 10 ETDRS Letters at Week 24: number analyzed (Participants) | 261 | 270
  Loss ≥ 10 ETDRS Letters at Week 24 | 17 | 12
  Loss ≥ 10 ETDRS Letters at Week 28: number analyzed (Participants) | 257 | 263
  Loss ≥ 10 ETDRS Letters at Week 28 | 21 | 14
  Loss ≥ 10 ETDRS Letters at Week 32: number analyzed (Participants) | 252 | 268
  Loss ≥ 10 ETDRS Letters at Week 32 | 23 | 16
  Loss ≥ 10 ETDRS Letters at Week 36: number analyzed (Participants) | 250 | 266
  Loss ≥ 10 ETDRS Letters at Week 36 | 22 | 18
  Loss ≥ 10 ETDRS Letters at Week 40: number analyzed (Participants) | 246 | 265
  Loss ≥ 10 ETDRS Letters at Week 40 | 21 | 24
  Loss ≥ 10 ETDRS Letters at Week 44: number analyzed (Participants) | 240 | 260
  Loss ≥ 10 ETDRS Letters at Week 44 | 18 | 21
  Loss ≥ 10 ETDRS Letters at Week 48: number analyzed (Participants) | 245 | 262
  Loss ≥ 10 ETDRS Letters at Week 48 | 24 | 25
  Loss ≥ 15 ETDRS Letters at Week 2: number analyzed (Participants) | 270 | 275
  Loss ≥ 15 ETDRS Letters at Week 2 | 3 | 4
  Loss ≥ 15 ETDRS Letters at Week 4: number analyzed (Participants) | 273 | 278
  Loss ≥ 15 ETDRS Letters at Week 4 | 4 | 4
  Loss ≥ 15 ETDRS Letters at Week 8: number analyzed (Participants) | 274 | 274
  Loss ≥ 15 ETDRS Letters at Week 8 | 4 | 4
  Loss ≥ 15 ETDRS Letters at Week 12: number analyzed (Participants) | 267 | 274
  Loss ≥ 15 ETDRS Letters at Week 12 | 6 | 3
  Loss ≥ 15 ETDRS Letters at Week 16: number analyzed (Participants) | 264 | 274
  Loss ≥ 15 ETDRS Letters at Week 16 | 9 | 5
  Loss ≥ 15 ETDRS Letters at Week 20: number analyzed (Participants) | 262 | 275
  Loss ≥ 15 ETDRS Letters at Week 20 | 7 | 6
  Loss ≥ 15 ETDRS Letters at Week 24: number analyzed (Participants) | 261 | 270
  Loss ≥ 15 ETDRS Letters at Week 24 | 7 | 6
  Loss ≥ 15 ETDRS Letters at Week 28: number analyzed (Participants) | 257 | 263
  Loss ≥ 15 ETDRS Letters at Week 28 | 7 | 5
  Loss ≥ 15 ETDRS Letters at Week 32: number analyzed (Participants) | 252 | 268
  Loss ≥ 15 ETDRS Letters at Week 32 | 10 | 9
  Loss ≥ 15 ETDRS Letters at Week 36: number analyzed (Participants) | 250 | 266
  Loss ≥ 15 ETDRS Letters at Week 36 | 14 | 9
  Loss ≥ 15 ETDRS Letters at Week 40: number analyzed (Participants) | 246 | 265
  Loss ≥ 15 ETDRS Letters at Week 40 | 18 | 13
  Loss ≥ 15 ETDRS Letters at Week 44: number analyzed (Participants) | 240 | 260
  Loss ≥ 15 ETDRS Letters at Week 44 | 8 | 11
  Loss ≥ 15 ETDRS Letters at Week 48: number analyzed (Participants) | 245 | 262
  Loss ≥ 15 ETDRS Letters at Week 48 | 15 | 13

5. Secondary Outcome: Proportion of Participants With BCVA Snellen Equivalent of 20/40 or Better Over Time (≥69 ETDRS Letters)
Description: as for outcome 1
Time Frame: Day 1 to Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Treatment Group A) | Aflibercept (Treatment Group B)
Number analyzed (Participants) | 276 | 281
Participants
  Snellen Equivalent of 20/40 or Better at Baseline | 122 | 129
  Snellen Equivalent of 20/40 or Better at Week 2: number analyzed (Participants) | 270 | 275
  Snellen Equivalent of 20/40 or Better at Week 2 | 148 | 152
  Snellen Equivalent of 20/40 or Better at Week 4: number analyzed (Participants) | 273 | 278
  Snellen Equivalent of 20/40 or Better at Week 4 | 156 | 165
  Snellen Equivalent of 20/40 or Better at Week 8: number analyzed (Participants) | 274 | 274
  Snellen Equivalent of 20/40 or Better at Week 8 | 156 | 165
  Snellen Equivalent of 20/40 or Better at Week 12: number analyzed (Participants) | 267 | 274
  Snellen Equivalent of 20/40 or Better at Week 12 | 148 | 171
  Snellen Equivalent of 20/40 or Better at Week 16: number analyzed (Participants) | 264 | 274
  Snellen Equivalent of 20/40 or Better at Week 16 | 149 | 172
  Snellen Equivalent of 20/40 or Better at Week 20: number analyzed (Participants) | 262 | 275
  Snellen Equivalent of 20/40 or Better at Week 20 | 151 | 179
  Snellen Equivalent of 20/40 or Better at Week 24: number analyzed (Participants) | 261 | 270
  Snellen Equivalent of 20/40 or Better at Week 24 | 158 | 183
  Snellen Equivalent of 20/40 or Better at Week 28: number analyzed (Participants) | 257 | 263
  Snellen Equivalent of 20/40 or Better at Week 28 | 151 | 175
  Snellen Equivalent of 20/40 or Better at Week 32: number analyzed (Participants) | 252 | 268
  Snellen Equivalent of 20/40 or Better at Week 32 | 147 | 174
  Snellen Equivalent of 20/40 or Better at Week 36: number analyzed (Participants) | 250 | 266
  Snellen Equivalent of 20/40 or Better at Week 36 | 147 | 179
  Snellen Equivalent of 20/40 or Better at Week 40: number analyzed (Participants) | 246 | 265
  Snellen Equivalent of 20/40 or Better at Week 40 | 151 | 174
  Snellen Equivalent of 20/40 or Better at Week 44: number analyzed (Participants) | 240 | 260
  Snellen Equivalent of 20/40 or Better at Week 44 | 149 | 178
  Snellen Equivalent of 20/40 or Better at Week 48: number analyzed (Participants) | 245 | 262
  Snellen Equivalent of 20/40 or Better at Week 48 | 144 | 175

6. Secondary Outcome: Proportion of Participants With BCVA Snellen Equivalent of 20/200 or Worse Over Time (≤38 ETDRS Letters)
Description: as for outcome 1
Time Frame: Day 1 to Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 (Treatment Group A) | Aflibercept (Treatment Group B)
Number analyzed (Participants) | 276 | 281
Participants
  Snellen Equivalent of 20/200 or Worse at Baseline | 17 | 15
  Snellen Equivalent of 20/200 or Worse at Week 2: number analyzed (Participants) | 270 | 275
  Snellen Equivalent of 20/200 or Worse at Week 2 | 11 | 12
  Snellen Equivalent of 20/200 or Worse at Week 4: number analyzed (Participants) | 273 | 278
  Snellen Equivalent of 20/200 or Worse at Week 4 | 10 | 14
  Snellen Equivalent of 20/200 or Worse at Week 8: number analyzed (Participants) | 274 | 274
  Snellen Equivalent of 20/200 or Worse at Week 8 | 11 | 13
  Snellen Equivalent of 20/200 or Worse at Week 12: number analyzed (Participants) | 267 | 274
  Snellen Equivalent of 20/200 or Worse at Week 12 | 11 | 12
  Snellen Equivalent of 20/200 or Worse at Week 16: number analyzed (Participants) | 264 | 274
  Snellen Equivalent of 20/200 or Worse at Week 16 | 11 | 10
  Snellen Equivalent of 20/200 or Worse at Week 20: number analyzed (Participants) | 262 | 275
  Snellen Equivalent of 20/200 or Worse at Week 20 | 13 | 13
  Snellen Equivalent of 20/200 or Worse at Week 24: number analyzed (Participants) | 261 | 270
  Snellen Equivalent of 20/200 or Worse at Week 24 | 11 | 13
  Snellen Equivalent of 20/200 or Worse at Week 28: number analyzed (Participants) | 257 | 263
  Snellen Equivalent of 20/200 or Worse at Week 28 | 12 | 13
  Snellen Equivalent of 20/200 or Worse at Week 32: number analyzed (Participants) | 252 | 268
  Snellen Equivalent of 20/200 or Worse at Week 32 | 14 | 18
  Snellen Equivalent of 20/200 or Worse at Week 36: number analyzed (Participants) | 250 | 266
  Snellen Equivalent of 20/200 or Worse at Week 36 | 14 | 13
  Snellen Equivalent of 20/200 or Worse at Week 40: number analyzed (Participants) | 246 | 265
  Snellen Equivalent of 20/200 or Worse at Week 40 | 14 | 17
  Snellen Equivalent of 20/200 or Worse at Week 44: number analyzed (Participants) | 240 | 260
  Snellen Equivalent of 20/200 or Worse at Week 44 | 9 | 15
  Snellen Equivalent of 20/200 or Worse at Week 48: number analyzed (Participants) | 245 | 262
  Snellen Equivalent of 20/200 or Worse at Week 48 | 15 | 15

7. Secondary Outcome: Mean Change in OCT Central Subfield Retinal Thickness (CST) From Baseline to the Average of Weeks 40, 44 and 48 and Over Time
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE) as assessed by a central reading center.
Time Frame: Day 1 to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | KSI-301 (Treatment Group A) | Aflibercept (Treatment Group B)
Number analyzed (Participants) | 276 | 281
Microns
  Week 2: number analyzed (Participants) | 270 | 274
  Week 2 | -72.1 (83.74) | -99.9 (93.75)
  Week 4: number analyzed (Participants) | 272 | 277
  Week 4 | -74.9 (98.33) | -109.4 (100.87)
  Week 8: number analyzed (Participants) | 274 | 274
  Week 8 | -89.1 (121.13) | -122.2 (109.58)
  Week 12: number analyzed (Participants) | 267 | 274
  Week 12 | -97.1 (118.62) | -126.3 (111.55)
  Week 16: number analyzed (Participants) | 266 | 274
  Week 16 | -107.2 (110.02) | -99.2 (110.47)
  Week 20: number analyzed (Participants) | 261 | 275
  Week 20 | -111 (112.97) | -125.5 (117.39)
  Week 24: number analyzed (Participants) | 262 | 270
  Week 24 | -109.9 (112.82) | -101.8 (113.21)
  Week 28: number analyzed (Participants) | 257 | 262
  Week 28 | -114.6 (111.47) | -124.1 (111.51)
  Week 32: number analyzed (Participants) | 251 | 268
  Week 32 | -111.9 (122.05) | -104.3 (116.09)
  Week 36: number analyzed (Participants) | 250 | 265
  Week 36 | -113.6 (129.84) | -124.4 (112.12)
  Week 40: number analyzed (Participants) | 246 | 265
  Week 40 | -113.6 (115.34) | -103.1 (109.25)
  Week 44: number analyzed (Participants) | 240 | 261
  Week 44 | -115.8 (115.81) | -129.4 (114.70)
  Week 48: number analyzed (Participants) | 245 | 262
  Week 48 | -117 (114) | -109.2 (120.75)
  Week 40-48 Average: number analyzed (Participants) | 253 | 268
  Week 40-48 Average | -114.6 (113.92) | -113.4 (112.07)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) reported through Week 52 or Early Termination (ET)
Arm/Group | KSI-301 (Treatment Group A) | Aflibercept (Treatment Group B)
All-Cause Mortality (participants affected / at risk) | 4/276 | 3/281
Serious Adverse Events (participants affected / at risk) | 39/276 | 39/281
Other Adverse Events (participants affected / at risk) | 110/276 | 80/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 (Treatment Group A) (N=276) | Aflibercept (Treatment Group B) (N=281)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Periorbital cellulitis - Study eye (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Retinal detachment - Study eye (Eye disorders) | 3 (3) | 0 (0)
Eye pain - Study eye (Eye disorders) | 1 (1) | 0 (0)
Uveitis - Study eye (Eye disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (2)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Intraocular pressure increased - Study eye (Investigations) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 (Treatment Group A) (N=276) | Aflibercept (Treatment Group B) (N=281)
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 22 (23) | 15 (16)
Vitreous floaters - Study eye (Eye disorders) | 21 (23) | 7 (7)
Conjunctival haemorrhage - Study eye (Eye disorders) | 20 (26) | 11 (17)
COVID-19 (Infections and infestations) | 34 (35) | 35 (35)
Urinary tract infection (Infections and infestations) | 15 (23) | 16 (21)
Hypertension (Vascular disorders) | 17 (17) | 14 (14)
Intraocular pressure increased - Study eye (Investigations) | 15 (17) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT04964089/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT04964089/SAP_001.pdf